CLINICAL TRIAL: NCT03563573
Title: Single-dose Potassium Supplementation in ADHD Patients With Lidocaine Ineffectiveness
Brief Title: Single-dose Potassium Supplementation in Patients With ADHD for Whom the Anesthetic Lidocaine is Ineffective
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: AlkaliDx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-01A
Record Dates: First submitted 2018-05-15; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: ADHD
Keywords: Conditions in which lidocaine is ineffective
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The trial will have 2 arms, lidocaine sensitive (effective) and lidocaine insensitive (ineffective). The sample will be enriched to have 50% in each arm. Within each arm, subjects will be randomized on a 1-to-1 allocation to the treatment or control groups.
  The investigators will adopt an iterative approach of testing of batches of subjects because (1) the frequency of lidocaine-insensitivity is only known approximately, (2) the frequency may be unevenly distributed across ethnic groups, and (3) the exact effect size of the potassium is not known, though reported to be high in off-label use in clinical settings with more chronic administration.
  At the end of testing 40 patients, the results will be analyzed for statistical significance. (1) If the results are statistically significant with a 95% confidence, the testing may stop with the first batch of 40 subjects. (2) If not, sequential, iterative batches of 20 subjects will be tested, and the results reanalyzed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The scoring of the lidocaine test is masked, using the coded identity of the tastes. The scoring will be done during the visit by the Scoring and Randomization Specialist so that the patient can be assigned to an intervention or control group to maintain equal numbers in treatment versus control groups. To prevent bias, the Scoring and Randomization Specialist will not be involved in any of the ADHD assessment steps and the patients will not be told about their lidocaine status until after all study testing is done. The subjects and other study personnel such as those doing the ADHD testing will be told not to discuss what they could or couldn't taste. Having scored the lidocaine test, the Scoring and Randomization Specialist will assign subjects to Intervention versus Control using a 1-to-1 allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lidocaine-effective ADHD: Intervention (Active Comparator): Single-dose potassium gluconate oral capsule intervention for ADHD subjects for whom lidocaine is effective
  Interventions: Drug: Potassium Gluconate Oral Capsule
- Lidocaine-effective ADHD: Placebo (Placebo Comparator): Single-dose placebo oral capsule intervention for ADHD subjects for whom lidocaine is effective
  Interventions: Drug: Placebo oral capsule
- Lidocaine-ineffective ADHD: Intervention (Active Comparator): Single-dose potassium gluconate oral capsule intervention for ADHD subjects for whom lidocaine is ineffective
  Interventions: Drug: Potassium Gluconate Oral Capsule
- Lidocaine-ineffective ADHD: placebo (Placebo Comparator): Single-dose placebo oral capsule intervention for ADHD subjects for whom lidocaine is ineffective
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Potassium Gluconate Oral Capsule — Each subject will receive a dose of ~8 mg/kg of potassium. We will be giving a maximum of 14 mEq in a single dose.
  Arms: Lidocaine-effective ADHD: Intervention; Lidocaine-ineffective ADHD: Intervention
Drug: Placebo oral capsule — Each subject will receive a dose of ~8 mg/kg of a placebo capsule
  Arms: Lidocaine-effective ADHD: Placebo; Lidocaine-ineffective ADHD: placebo

SUMMARY:
Randomized, controlled, double-blind trial of the effect of a single dose of potassium on ADHD symptoms as measured by changes in measures of symptoms of ADHD correlated with the results of their Lidocaine Effectiveness Test.

DETAILED DESCRIPTION:
Subjects with a confirmed diagnosis of Attention Deficit Hyperactivity Disorder (ADHD), who are either untreated or poorly controlled with existing ADHD therapy, will be recruited for a single, four-hour session.

Each subject will be tested for lidocaine effectiveness using the application of lidocaine gel to the tongue and assessment by taste.

The subjects will then be assigned to two arms, (1) lidocaine sensitive (effective) or (2) lidocaine insensitive (ineffective), and then randomized as to an intervention of potassium supplementation or a placebo.

Each subject will:

* Complete questionnaires about their history of certain symptoms and a food diary.
* Get an ECG to exclude those with arrhythmias.
* Have their baseline serum potassium tested
* Have measures of ADHD symptoms performed.

Then each subject will receive the intervention of a single dose of the potassium or placebo.

After the wait of one hour, a repeat serum potassium and measurement of symptoms will be performed.

Note; The FDA also requires a Columbia Suicide Severity Rating Scale (C-SSRS) for all ADHD trials

ELIGIBILITY:
Inclusion Criteria:

1. Previously documented ADHD diagnosis
2. Untreated or taking existing ADHD drugs, but symptoms poorly controlled (e.g., symptoms not well managed by amphetamines, including ongoing inattention and impulsivity)

Exclusion Criteria:

1. Well treated with existing ADHD medication
2. Epilepsy
3. IQ less than 80
4. Severe head trauma that led to loss of consciousness for more than an hour or required surgery
5. Birth weight below 5 pounds or 2270 grams
6. Severe autism (milder conditions described as Asperger syndrome or "high-functioning autism" are not excluded)
7. Comorbid psychiatric disorders, such as generalized anxiety disorder, major depressive disorder, schizophrenia and schizoaffective disorder, bipolar disorder, and any co-morbid condition at the discretion of the PI that would interfere with a patient's ability to participate
8. Mouth lesions, known to temporarily interfere with lidocaine effectiveness
9. Renal disease or abnormal kidney function or receiving dialysis
10. An individual has a factor likely to reduce penetrance, including excessive salt loss, such as caked salt on the body after exercise and Cystic fibrosis in a relative suggestive of the individual being a carrier.
11. Heart arrhythmia, known or evident on ECG
12. Known intolerance or allergy to lidocaine
13. Already taking supplemental potassium or renin angiotensin aldosterone inhibitors or other potassium elevating agents (see list below)

Angiotensin Converting Enzyme Inhibitors

1. Alacepril (not available in US)
2. Benazepril (Lotensin)
3. Captopril (trade name Capoten)
4. Cilazapril (Inhibace)
5. Delapril (not available in US)
6. Enalapril (Vasotec/Renitec)
7. Fosinopril (Fositen/Monopril)
8. Imidapril (Tanatril)
9. Lisinopril (Listril/Lopril/Novatec/Prinivil/Zestril)
10. Moexipril (Univasc)
11. Perindopril (Coversyl/Aceon/Perindo)
12. Quinapril (Accupril)
13. Ramipril (Altace/Prilace/Ramace/Ramiwin/Triatec/Tritace)
14. Spirapril (Renormax)
15. Temocapril (not available in US)
16. Teprotide (but not active by oral administration and not used in US)
17. Trandolapril (Mavik/Odrik/Gopten)
18. Zofenopril

Angiotensin receptor blockers

1. Azilsartan (Edarbi)
2. Candesartan (Atacand)
3. Eprosartan (Teveten)
4. Fimasartan (Kanarb)
5. Irbesartan (Avapro)
6. Losartan (Cozaar)
7. Olmesartan (Benicar/Olmetec)
8. Telmisartan (Micardis)
9. Valsartan (Diovan)

Aldosterone antagonists

1. Spironolactone (Aldactone)
2. Eplerenone (Inspra)

Renin inhibitors

a. Aliskiren (Tekturna, Rasilez)

Other potassium elevating agents

1. Antibiotics, including penicillin G and trimethoprim
2. Azole antifungals
3. Beta-blockers
4. Herbal supplements, including milkweed, lily of the valley, Siberian ginseng, Hawthorn berries
5. Heparin
6. Nonsteroidal anti-inflammatory medications (NSAIDs)
7. Oral contraceptives containing drospirenone

Ages: 13 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-11-04 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of lidocaine ineffectiveness in those with ADHD | Baseline
  Investigator assesses identification and intensity of tastes (such as sweet) before and after application of oral lidocaine gel to the tongue.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1-2 hours after intervention
  Investigator documentation of adverse reactions to either lidocaine or potassium
Other discomforts | 1-2 hours after intervention
  Investigator documentation of complaints or minor discomforts
Change in ADHD-RS questionnaires | Baseline and ~1-2 hours later, 1 hour after intervention
  The questionnaire is a standard assessment tool for measuring the level of ADHD symptoms. The ADHD-RS-IV is for adults and the ADHD-RSM-5 is for teenagers. This test has been validated for measuring the impact of drugs in ADHD, typically multi-dose, multi-week changes.
  Since this study is a single-dose, several-hour study, the Investigators will complete only the portions designed to done with the patient and by the clinician; sections designed to be completed by parents and teachers. The results will establish expectations for future multi-dose studies.
  All scores on a range of None, Mild, Moderate, Severe.
  1. Carelessness
  2. Difficulty sustaining attention in activities
  3. No follow through
  4. Can't organize
  5. Avoids/dislikes tasks requiring sustained mental effort
  6. Loses Important items
  7. Easily distractible
  8. Forgetful in daily activities
Change in Clinical Global Impression Physician Completed Questionnaire | Baseline and ~1-2 hours later, 1 hour after intervention
  Clinician-assessed improvement in overall symptoms, using CGI S (severity) as baseline and CGI I (improvement) to track any change.
  Investigator assesses "Compared to his or her condition at baseline, how much has he or she changed?"
  Very much improved Much improved Minimally improved No change Minimally worse Much worse Very much worse
Change in scores using Quotient ADHD System | Baseline and ~1 hour after intervention
  The Quotient device (http://www.quotient-adhd.com) tracks scores on 6 factors of motion analysis; 6 factors of attention response; and 8 factors of attention state. The subject plays a diagnostic "video game" and the machine tracks movement of the head, and speed and accuracy of the mouse clicks.
  The first assessment will serve as a baseline and the assessment post-intervention will measure any changes. (all scores from 0-100)
  Motion Analysis (including Immobility Duration, Number of movements, displacement, area, spacial complexity, temporal scaling)
  Attention Response Analysis (including adjusted Accuracy, Omission Errors, Commission Errors, Latency, Variability, Coefficient of Variation for response latency)
  Attention State Analysis (including number of shifts, Attentive, Impulsive, Distracted, Disengaged, Random, Minimal, Contrary, Overall Results)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Segal, MD PhD, Principal Investigator — PhenoSolve, LLC; Mark Mintz, MD, Principal Investigator — CNNH & CRCNJ
Locations (1):
- Clinical Research Center of New Jersey (CRCNJ), Voorhees Township, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to submit for publication descriptions of what was accomplished, and the evaluations as described in the study, including the incidence of lidocaine ineffectiveness in those with ADHD.
Supporting Information: CSR
Time Frame: When the study is complete
Access Criteria: open

REFERENCES:
- [Background] Infante MA, Moore EM, Nguyen TT, Fourligas N, Mattson SN, Riley EP. Objective assessment of ADHD core symptoms in children with heavy prenatal alcohol exposure. Physiol Behav. 2015 Sep 1;148:45-50. doi: 10.1016/j.physbeh.2014.10.014. Epub 2014 Oct 23. PMID 25447751
- [Background] Levitt JO. Practical aspects in the management of hypokalemic periodic paralysis. J Transl Med. 2008 Apr 21;6:18. doi: 10.1186/1479-5876-6-18. PMID 18426576
- [Background] Nakai Y, Milgrom P, Mancl L, Coldwell SE, Domoto PK, Ramsay DS. Effectiveness of local anesthesia in pediatric dental practice. J Am Dent Assoc. 2000 Dec;131(12):1699-705. doi: 10.14219/jada.archive.2000.0115. PMID 11143733
- [Background] Segal MM. We cannot say whether attention deficit hyperactivity disorder exists, but we can find its molecular mechanisms. Pediatr Neurol. 2014 Jul;51(1):15-6. doi: 10.1016/j.pediatrneurol.2014.04.014. Epub 2014 Apr 18. No abstract available. PMID 24938135
- [Background] Segal MM, Rogers GF, Needleman HL, Chapman CA. Hypokalemic sensory overstimulation. J Child Neurol. 2007 Dec;22(12):1408-10. doi: 10.1177/0883073807307095. PMID 18174562
- [Background] Segal MM, Douglas AF. Late sodium channel openings underlying epileptiform activity are preferentially diminished by the anticonvulsant phenytoin. J Neurophysiol. 1997 Jun;77(6):3021-34. doi: 10.1152/jn.1997.77.6.3021. PMID 9212254
- [Background] Teicher MH, Polcari A, Fourligas N, Vitaliano G, Navalta CP. Hyperactivity persists in male and female adults with ADHD and remains a highly discriminative feature of the disorder: a case-control study. BMC Psychiatry. 2012 Nov 7;12:190. doi: 10.1186/1471-244X-12-190. PMID 23134619
- See also: Rozanski RJ, Primosch RE, Courts FJ (1988). Clinical efficacy of 1 and 2% solutions of lidocaine. Pediatr Dent.10:287-90 — https://pdfs.semanticscholar.org/1778/f693dc7dd257ab98a96b5bf03408d9cef3eb.pdf
- See also: Saul R (2014) "ADHD Does Not Exist". HarperCollins. — https://www.amazon.com/ADHD-Does-Not-Exist-Hyperactivity/dp/006226673X
- See also: Segal MM, Jurkat-Rott K, Levitt J, Lehmann-Horn F (2014) Hypokalemic periodic paralysis - an owner's manual — http://simulconsult.com/resources/hypopp.html
- See also: Segal MM (2015) Devices, Kits, and Methods for Determining Sensitivity to Anesthetics. US Patent Filing 62/210,747, Filed 09/14/2015 — https://patents.google.com/patent/WO2017035470A1/en